CLINICAL TRIAL: NCT00915694
Title: A Phase I Trial of the Protease Inhibitor Nelfinavir and Concurrent Radiation and Temozolomide in Patients With WHO Grade IV Glioma
Brief Title: Nelfinavir Mesylate, Radiation Therapy, and Temozolomide in Treating Patients With Glioblastoma Multiforme
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000644278; UPCC-01309; IRB#809463
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult gliosarcoma; adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Nelfinavir; Temozolomide; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): NFV-RT-Tem
  Interventions: Drug: nelfinavir mesylate; Drug: temozolomide; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: nelfinavir mesylate
Drug: temozolomide
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Nelfinavir mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving nelfinavir mesylate together with radiation therapy and temozolomide may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of nelfinavir mesylate when given together with radiation therapy and temozolomide in treating patients with glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of nelfinavir mesylate when given concurrently with radiotherapy and temozolomide followed by temozolomide alone in patients with glioblastoma multiforme.
* Determine the safety and dose-limiting toxicities of this regimen in these patients.

Secondary

* Determine the progression-free survival (PFS) and overall survival (OS) of patients treated with this regimen.
* Compare the observed median values of PFS and OS obtained in this study to the historical median values of 6.9 months and 14.6 months, respectively.

OUTLINE: This is a dose-escalation study of nelfinavir mesylate.

Patients receive oral nelfinavir mesylate twice daily beginning 7-10 days before the initiation of chemoradiotherapy and continuing until the completion of chemoradiotherapy. Patients undergo radiotherapy once daily 5 days a week and receive concurrent oral temozolomide once daily for 6 weeks. Beginning 4 weeks after completion of nelfinavir mesylate and chemoradiotherapy, patients receive oral temozolomide alone once daily on days 1-5. Treatment with temozolomide repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed WHO grade IV supratentorial astrocytoma (glioblastoma multiforme)

  * Newly diagnosed disease
* Has undergone maximal surgical resection

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Serum creatinine < 1.5 times upper limit of normal (ULN)
* AST or ALT < 2 times ULN
* Serum bilirubin < 1.5 mg/dL
* No known HIV infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior cranial radiotherapy
* More than 30 days since prior investigational agents
* No other concurrent investigational agents
* No concurrent use of any of the following drugs:

  * Antiarrhythmics (i.e., amiodarone or quinidine)
  * Antimycobacterials (i.e., rifampin)
  * Ergot derivatives (i.e., dihydroergotamine, ergonovine, ergotamine, or methylergonovine)
  * Herbal products (i.e., St. John's wort)
  * HMG-CoA reductase inhibitors (i.e., lovastatin or simvastatin)
  * Neuroleptics (i.e., pimozide)
  * Sedatives and/or hypnotics (i.e., midazolam or triazolam)
* Concurrent corticosteroids allowed provided dose has been stable or decreasing for ≥ 14 days prior to study entry

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of nelfinavir mesylate | 90 days
Dose-limiting toxicities as assessed by NCI CTC v3.0 | 90 days

SECONDARY OUTCOMES:
Progression-free survival | One year
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jay F. Dorsey, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials